CLINICAL TRIAL: NCT00721695
Title: Randomized, Controlled, Double-Masked, Multicenter, Exploratory Study of the Clinical Benefit and Safety of OMS302 Injection in Subjects Undergoing Unilateral Cataract Extraction With Lens Replacement (CELR) Using a Coaxial Phacoemulsification Process
Brief Title: Exploratory Study of OMS302 Injection in Subjects Undergoing Unilateral Cataract Extraction by Phacoemulsification.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C07-005
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Cataract Extraction
Keywords: Cataract; Cataract Extraction; Lens Implantation; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): OMS302 Irrigation Solution
  Interventions: Drug: OMS302
- 2 (Active Comparator): OMS302-PE HCl Irrigation Solution
  Interventions: Drug: OMS302-PE
- 3 (Placebo Comparator): Standard topical mydriatics and BSS Irrigation Solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS302 — OMS302 Irrigation Solution
  Other Names: OMS302 Irrigation Solution
  Arms: 1
Drug: OMS302-PE — OMS302-PE HCI Irrigation Solution
  Other Names: OMS302-PE HCI Irrigation Solution
  Arms: 2
Drug: Vehicle — Standard topical mydriatics and Balanced Salt Solution Irrigation Solution
  Other Names: Standard topical mydriatics and Balanced Salt Solution Irrigation Solution
  Arms: 3

SUMMARY:
This is an exploratory study to determine the safety and clinical benefit of OMS302 Injection in subjects undergoing Cataract Extraction with Lens Replacement (CELR) using a coaxial phacoemulsification process.

DETAILED DESCRIPTION:
OMS302 Injection is a mydriatic/anti-inflammatory combination investigational drug product being developed as an irrigation solution during intracameral lens replacement surgical procedures of the eye. OMS302 irrigation solution may induce and maintain an adequately dilated pupil and reduce postoperative symptoms of discomfort such as eye pain and irritation. The use of OMS302 irrigation solution may eliminate the need for pre-operative dilation of the eye and could reduce the postoperative use of an anti-inflammatory and pain medications following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 50 years of age or older.
* Subject is to undergo unilateral primary CELR for an age-related cataract under topical anesthesia and using a clear cornea incision.
* Subject's history and physical examination are within normal limits or the examination is clinically non-significant for purposes of the study as determined by the Investigator, and subject is in good general health.
* Subject has best corrected visual acuity (BCVA) of 20/400 or better in the non-study eye.
* Subject has intraocular pressure (IOP) between 5 mmHg and 22 mmHg, inclusive, in the study eye.

Exclusion Criteria:

* Subject is allergic to any of the individual ingredients in OMS302
* Subject who is taking medications with the same activities as that of the active ingredients in OMS302 for defined time intervals prior to and after surgery.
* Female subject of childbearing potential (i.e., not surgically sterilized nor post-menopausal longer than one year) who is not using an effective method of birth control within at least 14 days prior to surgery or has a positive pregnancy test.
* Subject who has a present condition or history of any clinically significant uncontrolled gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, neurological, psychiatric, connective tissue, respiratory, or medical disorder as determined by the Investigator.
* Subject who is taking anticoagulants.
* Subject who is taking or needs to take for the duration of the study any of the prohibited medications.
* Subject with pseudo-capsular exfoliation, or evidence of prior iritis or of ocular trauma with iris damage, or who has used pilocarpine within six months of screening.
* Subject that has uncontrolled chronic ocular disease.
* Subject that has active corneal pathology or scarring noted in either eye (except superficial punctate keratopathy in the non-study eye).
* Subject that has extraocular/intraocular inflammation in either eye.
* Subject has an active bacterial and/or viral infection in either eye.
* Subject that has narrow-angle glaucoma, unstable glaucoma, or glaucoma being treated with prostaglandins or prostaglandin analogues.
* Subject taking, or has taken within the past year, an alpha adrenergic antagonist.
* Subject that has participated in or is currently participating in any investigational drug or device trial within the previous 30 days prior to the day of surgery.
* Subject that has had intraocular conventional surgery within the past three months or intraocular laser surgery within one month of the planned surgery in the study eye.
* Subject that requires the use of other topical medications during the trial except prophylactic antibiotics, topical lid care or glaucoma medications or tear replacement solutions.
* Subject that needs other ocular surgery at the time of the cataract extraction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pupil diameter | Day of Surgery
Pain and other measures of ocular discomfort | 14 days
Degree of inflammation in the anterior chamber | 14 days

SECONDARY OUTCOMES:
Ocular safety and changes in visual activity and intraocular pressure | 28 days
General measures of safety | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott Houston, Study Director — Omeros Corporation
Locations (4):
- United States (4):
  - Shasta Eye Medical Group, Redding, California
  - Chu Vision Institute, Bloomington, Minnesota
  - Silverstein Eye Centers, Kansas City, Missouri
  - Davis Duehr Dean, Madison, Wisconsin

REFERENCES:
- [Background] Behndig A, Eriksson A. Evaluation of surgical performance with intracameral mydriatics in phacoemulsification surgery. Acta Ophthalmol Scand. 2004 Apr;82(2):144-7. doi: 10.1111/j.1600-0420.2004.00241.x. PMID 15043530
- [Background] Lundberg B, Behndig A. Intracameral mydriatics in phacoemulsification cataract surgery. J Cataract Refract Surg. 2003 Dec;29(12):2366-71. doi: 10.1016/s0886-3350(03)00522-4. PMID 14709298